CLINICAL TRIAL: NCT06885801
Title: Evaluation of a Novel Nasal Conformer in Pediatric Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: East Tennessee Children's Hospital (Other)
Responsible Party: Principal Investigator, Justin Daggett, Principal Investigator, East Tennessee Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Device Feasibility
Other Study IDs: IRB-2025-069
Record Dates: First submitted 2025-03-12; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Cleft Lip; Nasal Surgical Procedures
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Standard first, anatomic second (Other): Patients are started with the standard nasal conformer for the first 3 months and then switched to the anatomic conformer for the second 3 months
  Interventions: Device: use of an anatomically designed nasal conformer
- Anatomic first, standard second (Other): Patients are started with the anatomic nasal conformer for the first 3 months and then switched to the standard conformer for the second 3 months
  Interventions: Device: use of an anatomically designed nasal conformer

INTERVENTIONS:
Device: use of an anatomically designed nasal conformer — this study will evaluate the use of a nasal conformer that has been designed to match the internal airway anatomy of the anterior nose rather than the standard hollow, conical conformer currently available on the market

SUMMARY:
This study compares the current commercially available nasal conformer available for use in cleft lip repair and nasal scar release to a novel, anatomically shaped conformer based upon typical nasal airspace shape. This will follow patients using both of these types of splints during the post-operative healing process with one group starting with the standard splint and then moving to the anatomic conformer and the second group beginning with the anatomic and them moving to the standard conformer. This study will evaluate the patient experience and outcomes of the 2 types of conformers, looking at the discomfort, device dislodgements, ease of use and occurrence of complications such as skin irritation and rashes or skin breakdown.

ELIGIBILITY:
Inclusion Criteria:

* Patient's undergoing primary cleft lip repair or release of nasal scarring

Exclusion Criteria:

* patient or parents declined participation postoperative nasal stenting is judged clinically inappropriate

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2030-06-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Ease of use | 6 months
  The patients or (parents for younger patients) will complete a questionnaire at the end of 3 months and 6 months after using each of the various types of conformer. These questionnaires will consist of a grading scale evaluating each of the conformer is a based on the ease of cleaning, inserting, and keeping the stent in place is evaluated
safety of the conformer | 6 months
  The patients or (parents of younger patients) will complete a questionnaire at the end of 3 months and 6 months after using each of the various types of conformer. The these will give them the opportunity to report the occurrence of adverse events such as skin rashes, skin irritation, skin breakdown, or stent breakage.